CLINICAL TRIAL: NCT01628744
Title: Autoantibodies Against Specific Cytokines in Adults With Severe Mycobacterial Infection
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: DMR-99-IRB-075-1
Record Dates: First submitted 2012-06-24; First posted 2012-06-27 (Estimated); Last update posted 2012-06-27 (Estimated); Status verified 2012-06

CONDITIONS: Mycobacterium Infection
MeSH Terms: conditions — Mycobacterium Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with mycobacterial infection

SUMMARY:
In adult, the prevalence of mycobacterial infections is increased with age is largely unknown. IFN-gamma-IL-12/23 axis or NF-kappaB pathways might also plays crucial roles in adult against mycobacteria. Based on this hypothesis, the investigators had applied a functional assay to these pathways in patients with mycobacterial infection.

ELIGIBILITY:
Inclusion Criteria:

* Patients with mycobacterial infection

Exclusion Criteria:

* Malignancy
* Severe autoimmune
* HIV infection

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Pateitns with Mycobacterium, Particular to the non Tuberculosis mycobacterium infection, in Taiwan
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2011-01; Study Completion 2014-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Cheng-Lung KU, Ph.D, Principal Investigator — Graduate Institute of clinical Medical Science, China Medical Univerity, Taiwan
Locations (1):
- Graduate Institute of Clinical Medical Science, China Medical University, Taichung, Taiwan